CLINICAL TRIAL: NCT02059720
Title: Haplo-mismatch Donor Stem Cell Transplantation (SCT) Versus Autologous SCT Followed or Not by Maintenance Therapy, for Patients With Acute Myeloid Leukemia (AML) in First Remission: A Chinese Randomized Multicenter Study
Brief Title: Haplo-SCT vs ASCT With or Without Decitabine in AML CR1
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Collaborators: European Society for Blood and Marrow Transplantation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SZ3702; ChiCTR-TRC-14004196 (Registry Identifier: Chinese Clinical Trial Registry (ChiCTR))
Record Dates: First submitted 2014-02-10; First posted 2014-02-11 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Acute Myeloid Leukemia
Keywords: acute myeloid leukemia; allogeneic hematopoietic stem cell transplantation; autologous hematopoietic stem cell transplantation; maintenance treatment; hematopoietic stem cell transplantation
MeSH Terms: conditions — Leukemia, Myeloid, Acute

ARMS (2):
- auto (Active Comparator): patients receive autologous SCT
  Interventions: Procedure: HSCT
- haplo (Active Comparator): patients receive haplo-SCT
  Interventions: Procedure: HSCT

INTERVENTIONS:
Procedure: HSCT — Patients randomly assigned in to either of groups will receive either autologous SCT or haplo-SCT after CR1 is achieved.

SUMMARY:
A multicentre, prospective, open-label clinical study, including a randomized controlled study in low or intermediate-risk group patients, and a cohort study of maintenance treatment with decitabine after ASCT.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18y
* Diagnosed as AML (except acute promyelocytic leukemia M3) for the first time
* Minimal Residual Disease (MRD) test can be achieved (molecular biology first if applicatable, and/or cytogenetics and/or immunophenotyping)
* Presence of an available haplo-mismatch related donor

Exclusion Criteria:

* Contra-indications of chemotherapy or hematopoietic stem cell transplantation
* Presence of an available identical sibling donor or a 10/10 HLA loci-matched unrelated donor
* Participating in other clinical trials concerning the prophylaxis of disease recurrence after ASCT
* No effective contraception
* Pregnant or lactating females
* Other causes which are not suitable for the trial in investigator's consideration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2014-02; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Leukemia-Free Survival | Five years
  Defined as the survival duration starting at the day of graft infusion, terminating at the day of death, morphological relapse or the end of follow-up.

SECONDARY OUTCOMES:
Overall survival | Five years
  Defined as the survival duration starting at the day of graft infusion, terminating at the day of death or the end of follow-up.
Cumulative relapse incidence | Five years
  Defined as the cumulative incidence of morphological relapse after the day of graft infusion.
Non-relapse Mortality | Five years
  Defined as the cumulative incidence of death without cause of disease recurrence, which include the cause of GVHD, infection, hemorrhage, organic function failure, etc.
Cumulative incidence of engraftment | 180 days
  Defined as the cumulative incidence of durable complete donor chimerism detected by STR-PCR.

OTHER OUTCOMES:
Quality of Life | Five years
  Including incidence and severity of acute and chronic GVHD, activity of daily living, psychological status, recovery of professional activity, social adaption, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Depei Wu, M.D., Ph.D., Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The Fisrt Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China